CLINICAL TRIAL: NCT01876095
Title: Discontinuing Inappropriate Medication in Nursing Home Residents (the DIM NHR Study): a Cluster Randomized Controlled Trial
Brief Title: Discontinuing Inappropriate Medication in Nursing Home Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Katja Taxis, Professor of Pharmacotherapy and Clinical Pharmacy, University of Groningen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DIM-NHR study
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Polypharmacy Because of Multimorbidity in Geriatric Nursing Home Residents

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multidisciplinary medication review (Experimental): The multidisciplinary medication review consists of 5 steps:
  Step #1: Assessing patients' experiences and preferences regarding medicine use en assessing their medical history, allergies and lab results Step #2: Drug reviewing to assess contra-indicated medication and duplicate medication using consensus criteria e.g. START STOPP Beers criteria Step #3: Reflecting on results of drug reviewing Step #4: Setting up a pharmacotherapeutical action plan Step #5: Execution of pharmacotherapeutical action plan
  Interventions: Procedure: Multidisciplinary medication review
- usual care (No Intervention): Includes medication safety monitoring and ad hoc medication reviews on clinical indication that differ in quality and frequency, but no standardized multidisciplinary multistep medication reviews in the way as described for the intervention arm

INTERVENTIONS:
Procedure: Multidisciplinary medication review — Consists of the following steps:
  * 1. Elderly care physician and nursing staff evaluate with the patient the experience of taking medicines, adverse drug reactions and patient's preferences.
  * 2. Pharmacist reviews medication to identify drug related problems using START/STOPP en Beers criteria.
  * 3/4. Meeting of elderly care physician, pharmacist. Possibilities to discontinue prescribed medication will be examined resulting in pharmaceutical care plan that optimizes the patient's medication i.e. which inappropriate medication should be discontinued following a prioritization and time schedule.
  * 5. Execution of pharmaceutical care plan according to agreed schedule.
  Arms: Multidisciplinary medication review

SUMMARY:
Nursing home residents are among the frailest patient groups with a high number of co-morbidities and a high use of medicines. Inappropriate polypharmacy (i.e. often overprescribing) is one of the major problems in the nursing home population increasing the number of adverse drug reactions, falls, hospital admissions, mortality as well as having an impact on health care utilization. Multidisciplinary medication reviews have a great potential to reduce inappropriate medication use. The purpose of this study is to determine the efficacy of a multidisciplinary medication review model focussing on discontinuing inappropriate medication in a cluster randomized controlled trial in 600 nursing home residents. The primary outcome measure is the difference in proportion of residents who successfully discontinued medication between intervention and control group after four months. Secondary outcome measures will be the drug burden index, adverse drug withdrawal events related to the discontinued medication, death, referral to hospitals and quality of life.

ELIGIBILITY:
Nursing Home Wards:

Inclusion criteria:

* Long stay ward
* Capability and commitment to perform a multidisciplinary multistep medication review.

Exclusion criteria:

* Short stay, revalidation or observation wards
* Specialized ward where patients with an atypical etiology are cared for.
* Elderly care physicians who have recently received or who are to receive recertification at short notice with regard to systematic medication review methodology.
* Participation in other studies aimed at improving the quality of drug prescription (in the past 12 months).

Nursing Home Residents:

Inclusion criteria:

* A life expectancy of >4 weeks as judged by the treating elderly care physician.
* IC provided by patients themselves or provided by a legal representative for incapacitated patients.

Exclusion criteria:

* Refusal of treatment with medicines.
* Having received a multidisciplinary systematic medication review in the past 6 months.
* Being terminally ill and having a life expectancy ≤ 4 weeks as judged by the treating elderly care physician.
* Other reasons at the discretion of the elderly care physician / nursing staff

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 992 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Successful medication discontinuation | 4 months
  The number of residents for whom ≥1 inappropriate medication(s) are succesfully discontinued i.e. without relapse or severe withdrawal effects

SECONDARY OUTCOMES:
Medication initiation | 4 months
  Number of residents for whom ≥1 medication(s) are initiated (s) that should be started on the basis of the Screening Tool to Alert doctors to Right Treatment (START) criteria
Dose adjustment | 4 months
  Number of residents for whom ≥1 dose(s) are lowered or increased
Safer alternative medication | 4 months
  The percentage of residents for whom ≥1 medication(s) is replaced by a safer alternative
Drug burden index | 4 months
  A measure of a person's cumulative exposure to anticholinergic and sedative medications, which has been associated with falls in nursing home patients
Quality of Life | 4 months
  Quality of life will be measured using a disease specific instrument (DQI (Scholzel-Dorenbosch et al, in press) and a generic instrument EQ-5D-5L for all patients (Herdman et al, 2011).
adverse drug withdrawal events | 4 months
  The rate of adverse drug withdrawal events related to the discontinued medication
Death | 4 months
  Incidence of death
Hospital admission | 4 months
  Hospital admission
Falling | 4 months
  Defined as any event in which a nursing home resident touches the ground in an unintentional sudden manner without cues of emergency
Bone fractures | 4 months
  Bone fractures caused by falling
number of visits to outpatient clinics / emergency rooms / by medical consultants | 4 months
  number of visits to outpatient clinics, emergency rooms, number of visits by medical consultants i.e. physicians who visit the patients in the nursing homes,

OTHER OUTCOMES:
Cognitive function | 4 months
  Cognitive function as assessed with standardized cognitive tests called the Severe Impairment Battery and the Mini Mental Status Examination
Neuropsychiatric Symptoms | 4 months
  Assessment of change in neuropsychiatric symptoms (e.g. hallucinations & delusions) with the Neuropsychiatric Inventory (NPI) (nursing home version).

CONTACTS AND LOCATIONS:
Overall Officials: Katja Taxis, PhD, Principal Investigator — Groningen University
Locations (1):
- University of Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Wouters H, Scheper J, Koning H, Brouwer C, Twisk JW, van der Meer H, Boersma F, Zuidema SU, Taxis K. Discontinuing Inappropriate Medication Use in Nursing Home Residents: A Cluster Randomized Controlled Trial. Ann Intern Med. 2017 Nov 7;167(9):609-617. doi: 10.7326/M16-2729. Epub 2017 Oct 10. PMID 29052691
- [Derived] Wouters H, Quik EH, Boersma F, Nygard P, Bosman J, Bottger WM, Mulder H, Maring JG, Wijma-Vos L, Beerden T, van Doormaal J, Postma MJ, Zuidema SU, Taxis K. Discontinuing inappropriate medication in nursing home residents (DIM-NHR Study): protocol of a cluster randomised controlled trial. BMJ Open. 2014 Oct 8;4(10):e006082. doi: 10.1136/bmjopen-2014-006082. PMID 25296655